CLINICAL TRIAL: NCT06786078
Title: PREVAIL: a Clinical Investigation on Providing Reduced Effects of Visible Alopecia Caused by Chemotherapy Using the Lily Device - a Safety and Efficacy Study.
Brief Title: The Lily Device Trial
Acronym: PREVAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luminate Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLIN-1
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Chemotherapy Induced Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: Lily Device

INTERVENTIONS:
Device: Lily Device — Participants will wear the Lily Device at each chemotherapy session for the prescribed duration, where the device must be used during infusion and for at least two (2) hours and up to four (4) hours post infusion.

SUMMARY:
The goal of this clinical trial is to test if the Lily Device works to reduce chemotherapy induced hair loss in patients. It will also learn about the safety of the Lily Device. The main questions it aims to answer is:

* Do patient preserve their hair using the Lily Device after 4 cycles of chemotherapy, when hair preservation is a Grade ≤1 graded by an independent healthcare professional on the Common Terminology Criteria for Adverse Events (CTCAE)?
* What is the subject incidence of Grade 1 or above Adverse Device Events (ADE's)?

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ age 18 with breast cancer stage 1, 2 or 3, who have been deemed appropriate for (neo-)adjuvant chemotherapy and have not yet begun any systemic therapy.
2. Planned intravenous chemotherapy in the adjuvant or neoadjuvant setting with at least 4 cycles of chemotherapy, with one of the following regimens:

   * Doxorubicin 60 mg/m^2 with cyclophosphamide 600 mg/m^2 every 2-3 weeks
   * Doxorubicin 60 mg/m^2 with fluorouracil 500 mg/m^2 and cyclophosphamide 500 mg/m^2 every 2-3 weeks
   * Paclitaxel 80-90 mg/m^2 weekly (every 3 weeks constitutes a cycle)
   * Paclitaxel 175 mg/m^2 every 2-3 weeks
   * Paclitaxel 80-90 mg/m^2 weekly (every 3 weeks constitutes a cycle) with carboplatin AUC 1.5 every week
   * Paclitaxel 80-90 mg/m^2 weekly (every 3 weeks constitutes a cycle) with carboplatin AUC 5-6 every 3 weeks
   * Docetaxel 75-100 mg/m^2 every 3 weeks
   * Docetaxel 75 mg/m^2 with cyclophosphamide 600 mg/m^2 every 3 weeks
   * Docetaxel 75 mg/m^2 with carboplatin AUC 5-6 every 3 weeks

     * Concurrent administration with targeted agents/immunotherapy at standard doses (such as trastuzumab, pertuzumab, pembrolizumab) is allowed. Duration of targeted agents/immunotherapy is at the investigator's discretion.
     * Participants on AC-T regimens who are prescribed with at least 4 treatments with anthracycline followed by at least 4 treatments with taxane are eligible for the study. In terms of data analysis, these participants are counted towards the anthracycline group
3. Head size within the specified study sizing range.
4. Plan to complete chemotherapy in ≤ 12 months.
5. Willing and able to sign informed consent.
6. Willing to comply and tolerate all study procedures including:

   * Wearing the Lily device for the prescribed duration (device to be fitted before chemotherapy infusion, and worn during infusion and for at least two (2) hours and up to four (4) hours post infusion),
   * Complete all study related questionnaires.
   * Having photographs taken of the head at each visit.

To note:

* Participants who experience a hypersensitivity reaction to chemotherapy are allowed to continue in the study if the standard doses are maintained.
* Participants on the chemotherapy plan KEYNOTE-522 are eligible for this study.
* If a participant is prescribed a different chemotherapy treatment plan, they may be eligible for the study only if prior Sponsor approval is obtained.

Exclusion Criteria:

1. Baseline alopecia defined as CTCAE v5.0 grade > 0.
2. History of autoimmune disease associated with hair loss, e.g., alopecia areata, systemic lupus.
3. History of whole brain irradiation.
4. Recent chemotherapy (≤ 2 years), which caused hair loss.
5. Participants who are receiving or are planning to receive hormone replacement therapy or anti-estrogen therapy during the study, whereby the therapy in question has a known profile for causing hair loss.
6. Prescribed chemotherapy regimen with concurrent administration of taxane-based and anthracycline-based chemotherapy (i.e., infusion of both taxane and anthracycline agents on the same day).
7. Positive pregnancy test at baseline for participants with childbearing potential, as per standard of care for chemotherapy patient.
8. Known or suspected allergy or hypersensitivity to any component of the Lily device that comes into contact with the study participant.
9. Participants with a history of Temporomandibular Joint Disorder.
10. Any open wounds or sores on the participant's scalp or on part of the face where the device will be applied, which in the opinion of the investigator will not be healed prior to chemotherapy commencing.
11. Serious infection or medical illness which would jeopardize the ability of the participant to complete the planned chemotherapy.
12. Intercurrent life-threatening malignancy.
13. An existing history of scalp metastases or suspicion of presence of scalp metastasis.
14. Use of a cold cap, scalp cooling device or any other hair loss reduction device during the study.
15. Participants who, in the opinion of the investigator, will be inappropriate for inclusion into this study or will not comply with requirements of the study.
16. Participants who do not have the mental or physical ability to comply with time schedules and further study procedures.
17. Current participation in a clinical study or within the last 30 days prior to screening that may cause hair loss.
18. Participation in this study at an earlier stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Success in hair preservation using the Lily device after 4 cycles of chemotherapy, where hair preservation is defined as CTCAE v5.0 grade ≤ 1 alopecia determined by an independent healthcare professional. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
  A cycle of chemotherapy relates to the delivery of the chemotherapy regimen. In particular:
  * Participants on regimens delivered every 3 weeks - 1 chemotherapy treatment = 1 cycle.
  * Participants on regimens delivered every 2 weeks - 1 chemotherapy treatment = 1 cycle.
  * Participants on regimens delivered every 1 week - 3 chemotherapy treatments = 1 cycle.
  In CTCAE v5.0 alopecia grades are described as below:
  * Grade 0: No hair loss
  * Grade 1: Hair loss of <50% of normal for that individual that is not obvious from a distance but only on close inspection; a different hair style may be required to cover the hair loss, but it does not require a wig or hair piece to camouflage.
  * Grade 2: Hair loss of ≥50% normal for that individual that is readily apparent to others; a wig or hair piece is necessary if the patient desires to completely camouflage the hair loss; associated with psychosocial impact.
Primary Safety Endpoint - Subject incidence of Grade 1 or above ADE, graded with Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | From enrollment in the study until the end of study visit, taking place 30 days after the last treatment visit
  Adverse events will be graded as per the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Hair preservation experienced with the Lily device after 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)as assessed by the Subject according to the Dean Scale, with Grade 0, 1 or 2 defined as success. | After 4 cycles of chemotherapy
  A cycle of chemotherapy relates to the delivery of the chemotherapy regimen. In particular: - Participants on regimens delivered every 3 weeks - 1 chemotherapy treatment = 1 cycle. - Participants on regimens delivered every 2 weeks - 1 chemotherapy treatment = 1 cycle. - Participants on regimens delivered every 1 week - 3 chemotherapy treatments = 1 cycle.
  In the Dean Scale alopecia grades are described as below:
  * Grade 0: No hair loss
  * Grade 1: Hair loss of <25%
  * Grade 2: Hair loss of 25% ≤ hair loss < 50%
  * Grade 3: 50% ≤ hair loss < 75%
  * Grade 4: hair loss ≥ 75%
Concordance between percentage of patients with hair preservation after 4 cycles of chemotherapy as assessed by the independent healthcare professional and by the Subject. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Percentage of patients with success in hair preservation using the Lily device after 4 cycles of chemotherapy in subgroups of Subject race. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Percentage of patients with success in hair preservation using the Lily device after 4 cycles of chemotherapy in subgroups of Subject ethnicity. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Percentage of patients with success in hair preservation using the Lily device after 4 cycles of chemotherapy in subgroups of chemotherapy regimens. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Percentage of patients with success in hair preservation using the Lily device after 4 cycles of chemotherapy in subgroups of study site. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Quality of life experienced by the Subject as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) quality-of-life metrics after 4 cycles of chemotherapy. | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Compliance rate, defined as the ratio of prescribed wear time versus actual wear time. | From enrollment to the end treatment at the last cycle (each cycle is 14 - 21 days dependent on the chemotherapy regimen)
Event incidence of Grade 1 or above ADE. | From study enrollment to the end of study visit, 30 days after the last treatment visit (i.e 30 days after their final chemotherapy treatment and final treatment with the Lily Device)
Subject incidence of ADEs by grade, as measured with CTCAE v5.0. | From enrollment to the end of study visit, 30 days after the last treatment visit (i.e 30 days after their final chemotherapy treatment and final treatment with the Lily Device)
Subject incidence of serious ADEs. | From enrollment to the end of study visit, 30 days after the last treatment visit (i.e 30 days after their final chemotherapy treatment and final treatment with the Lily Device).
Adverse events of special interest (AESIs) incidence relating to scalp metastasis. | From enrollment to the end of study visit, 30 days after the last treatment visit (i.e 30 days after their final chemotherapy treatment and final treatment with the Lily Device).

OTHER OUTCOMES:
Percentage of patients with hair preservation by hair type, based on standardized photographs acquired as part of the primary endpoint | After 4 cycles of chemotherapy (each cycle is 14 - 21 days dependent on the chemotherapy regimen)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Inspira Health - Mullica Hills, Mullica Hill, New Jersey
  - Inspire Health - Vineland, Vineland, New Jersey
  - Guthrie - Our Lady of Lourdes Memorial Hospital, Binghamton, New York
  - Clinical Research Alliance, Westbury, New York
  - Guthrie Sayer Medical Centre, Sayre, Pennsylvania